CLINICAL TRIAL: NCT03339401
Title: Study to Assess the Safety, Overall Tolerability, and Antiviral Activity of Brincidofovir Versus Standard of Care for Treatment of Adenovirus in High-risk Pediatric Allogeneic Hematopoietic Transplant Recipients
Brief Title: The AdAPT Trial; Adenovirus After Allogeneic Pediatric Transplantation
Acronym: AdAPT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated due to low enrollment rate
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMX001-999
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Adenovirus
Keywords: Adenovirus; Pediatric; Hematopoietic Cell Transplant; Brincidofovir; Standard of care
MeSH Terms: conditions — Adenoviridae Infections | interventions — Standard of Care; brincidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brincidofovir (Experimental): Brincidofovir (BCV) for the treatment of adenovirs (AdV) infection in high-risk pediatric allogeneic hematopoietic cell transplant (HCT) recipients.
  Brincidofovir (BCV) treatment began no later than 100 days post-transplant and was to continue for a maximum of 16 weeks. Brincidofovir (BCV) was discontinued once AdV viremia was confirmed undetectable.
  Subjects who did NOT receive concurrent cyclosporine on Day 1:
  * If ≥48kg body weight, one 100mg oral tablet BIW (or 10mL of 10mg/mL oral suspension if unable to take tablets).
  * If <48kg body weight, 2mg/kg oral volume of 10mg/mL oral suspension BIW.
  Subjects who received cyclosporine on Day 1 (or initiated cyclosporine at any time):
  * 1.4mg/kg (maximum of 70mg) oral volume of 10mg/mL oral suspension BIW.
  * 2mg/kg (maximum of 100mg) oral volume of 10mg/mL oral suspension BIW if discontinued cyclosporine.
  Interventions: Drug: Brincidofovir
- Standard of Care (Other): Local institutional standard of care (SoC) (i.e., investigator-assigned therapy) for the treatment of adenovirus infection in high-risk pediatric allogeneic hematopoietic cell transplant (HCT) recipients.
  Management of these subjects was prescribed by the investigator as being in the best interests of the subject and may have included a "watch-and-wait" approach, with or without decreased immunosuppression (ergo, no treatment), or treatment administration with other available antivirals, most commonly cidofovir intravenously.
  Decisions regarding SoC, including administration of therapy, dose and regimen of therapy, modification of immunosuppression, and monitoring was the responsibility of the clinical team caring for the subject, according to institutional guidelines, local practices, and applicable guidelines for the management of AdV infection.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Local institutional standard of care (SoC) (i.e., investigator-assigned therapy) for the treatment of adenovirus infection in high-risk pediatric allogeneic hematopoietic cell transplant (HCT) recipients.
  Other Names: SoC
  Arms: Standard of Care
Drug: Brincidofovir — Brincidofovir (BCV) for the treatment of adenovirus infection in high-risk pediatric allogeneic hematopoietic cell transplant (HCT) recipients.
  Other Names: BCV
  Arms: Brincidofovir

SUMMARY:
This study was designed to assess the safety, overall tolerability, and antiviral activity of "short course" brincidofovir (BCV) therapy, as compared with current standard of care (SoC), for the treatment of adenovirus (AdV) infections in high-risk (i.e., T cell depleted) pediatric allogeneic hematopoietic cell transplant (HCT) recipients. A virologic response-driven approach to the duration of treatment was to be evaluated, in which subjects randomized to BCV therapy were to be treated until AdV viremia was confirmed as undetectable or until a maximum of 16 weeks of therapy, whichever occurred first. The formulation of BCV used in this study was oral tablet/suspension.

DETAILED DESCRIPTION:
This was a randomized, open-label, multi-center study of the safety, overall tolerability, and antiviral activity of BCV, as compared with SoC, in pediatric (and young adults in the United States) recipients of high-risk (i.e., T cell-depleted and/or unrelated cord blood graft, or a T cell-replete graft from ahaploidentical donor with post-transplant cyclophosphamide administration) allogeneic HCT. Subjects with AdV detected in plasma after their qualifying transplant could be screened for participation in the study. Subjects who met all applicable entry criteria were randomized in a 2:1 ratio to receive either BCV or SoC (i.e., investigator-assigned therapy). The formulation of BCV used in this study was oral tablet/suspension. Subjects were randomized within 100 days post-transplant; for study purposes, the day of randomization was defined as Day 1. During randomization, subjects were stratified based on the following variables: last AdV viremia (≥10,000 copies/mL versus <10,000 copies/mL) measurement available from the designated central virology laboratory prior to randomization, time from transplant to randomization (≥28 days versus <28 days), and T cell-depletion methodology (receipt of alemtuzumab or ex vivo depletion versus receipt of anti-thymocyte globulin [ATG] or no T cell depletion).

ELIGIBILITY:
Inclusion Criteria:

Subjects were high-risk allogeneic hematopoietic cell transplant (HCT) recipients aged 2 months to <18 years (<26 years in the United States) who met adenovirus (AdV) viremia criteria within 7 days of randomization (Day 1), and all other eligibility criteria. High-risk was defined as having received 1 of the following:

* A T cell-depleted graft:

  * Ex vivo T cell depletion via positive selective (e.g., CD34+ cell) or negative selection (e.g., T cell receptor α/β or CD3+ cell removal by column filtration); or
  * Serotherapy with ATG (cumulative dose of ≥3 mg/kg rabbit-derived ATG or ≥30 mg/kg of equine-derived ATG) administered within 10 days prior to transplant or at any time post-transplant and prior to Day 1; or
  * Serotherapy with alemtuzumab administered within 30 days prior to transplant or at any time post-transplant and prior to Day 1; or
* A cord blood graft from an unrelated donor with or without T cell depletion, or
* A T cell-replete graft from a haploidentical donor with high-dose cyclophosphamide (e.g., cumulative dose of ≥100 mg/kg) administered at any time post-transplant and prior to Day 1.

Subjects must have had qualifying AdV viremia within 100 days of transplant, which was defined as having either:

1. Confirmed AdV viremia of ≥1000 copies/mL on 2 consecutive AdV DNA polymerase chain reaction (PCR) test results drawn ≥48 hours apart from the designated central virology laboratory, with the second result being greater than the first; or
2. A single AdV viremia result of ≥10,000 copies/mL from the designated central virology laboratory Subjects who were previously treated with intravenous (IV) cidofovir (CDV) could have a cumulative exposure to IV CDV of no more than 10 mg/kg within 21 days prior to Day 1.

Written informed consent (and assent, where applicable) to participate in the study was obtained from each subject and his/her legal guardian(s) in accordance with national or local law and institutional practice.

Exclusion Criteria:

1. Any United States National Institutes of Health (NIH)/National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 4 diarrhea (i.e., life-threatening consequences with urgent intervention indicated) within 7 days prior to Day 1.
2. Any CTCAE Grade 2 or 3 diarrhea (i.e., increase of ≥4 stools/day over baseline [pre-transplant] diarrheal output), unless attributed to AdV, within 7 days prior to Day 1.
3. NIH Stage 4 acute graft versus host disease (GVHD) of the skin (i.e., generalized erythroderma with bullous formation) within 7 days prior to Day 1.
4. NIH Stage ≥2 acute GVHD of the liver (i.e., bilirubin >3 mg/dL [SI: >51 µmol/L]) within 7 days prior to Day 1.
5. NIH Stage ≥2 acute GVHD of the gut (i.e., diarrhea >556 mL/m2/day for pediatric patients [or >1000 mL/day for young adults at centers in the United States only], or severe abdominal pain with or without ileus) within 7 days prior to Day 1.
6. Poor clinical prognosis (including active malignancy or use of vasopressors other than low dose (e.g., ≤5 µg/kg/min) dopamine for renal perfusion within 7 days prior to Day 1.
7. Requirement for mechanical ventilation within 7 days prior to Day 1 or requirement for sustained oxygen delivery for >24 hours within 7 days prior to Day 1.
8. Concurrent HIV, active hepatitis B virus, or hepatitis C virus infection.
9. Specified out of range laboratory results (including alanine aminotransferase >5x the upper limit of normal [ULN], aspartate aminotransferase >5x ULN, total bilirubin >3 mg/dL [SI: >51 µmol/L], or prothrombin time-international normalized ratio >2x ULN) within 7 days prior to Day 1.
10. Estimated creatinine clearance <30 mL/min or use of renal replacement therapy within 7 days prior to Day 1.
11. Previous receipt of BCV at any time or receipt of CDV (IV or intravesicular) or letermovir within 48 hours prior to Day 1.
12. Received any anti-AdV-specific cell-based therapy within 6 weeks prior to Day 1 or previously received an anti-AdV vaccine at any time.

When applicable, female subjects of childbearing potential (i.e., not pre-menarche) were not pregnant or breastfeeding, and if sexually active, agreed to use 2 acceptable forms of contraception, 1 of which must have been a barrier method and the other a highly-effective method of contraception. Male subjects, if sexually active and capable of fathering a child, agreed to use a barrier method of contraception while enrolled in the study and for at least 90 days after the last dose of BCV.

Ages: 2 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (11):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Chicago, Chicago, Illinois
  - Joseph M. Sanzari Childrens Hospital-Regional Cancer Care, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Washington-Seattle Childrens Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (3):
  - IHOPe-Institut d'Homatologie et d'Oncologie Pediatrique, Lyon
  - Hopital Necker-Enfants Malades, Paris
  - Hopital Universitaire Robert Debre, Paris
- Germany (3):
  - Universitatsklinik fur Kinder-und Jugendmedizin, Tübingen, Baden-Wurttemberg
  - Dr. von Haunersches Kinderspital, Abteilung fur Padiatrische, München, Bavaria
  - Charite Universitatsmedizin Berlin, Campus Virchow-Klinikum, Berlin
- Our Lady's Children Hospital, Dublin, Ireland
- Italy (2):
  - Fondazione MBBM-CTMO Pediatrico, Monza
  - Ospedale Pediatrico Bambino Gesu, Roma
- Netherlands (2):
  - Leiden University Medical Center (LUMC), Leiden
  - Princess Maxima Center Utrecht, Utrecht
- Uniwerstytecki Azpital Kliniczny we Wroclawiu, Wroclaw, Lower Silesian Voivodeship, Poland
- Spain (2):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
- United Kingdom (11):
  - Royal Marsden Hospital, Sutton, Surrey
  - Newcastle-upon-Tyne Hospitals-Great Childrens Hospital, Newcastle upon Tyne, Tyneside
  - Birmingham Childrens Hospital, Birmingham, West Midlands
  - Leeds Children's Hospital, Leeds, West Yorkshire
  - Bristol Royal Hospital for Children, Bristol
  - Royal Hospital for Sick Children, Glasgow
  - University College London Hospital, London
  - St Marys Hospital, London
  - Great Ormond Street Hospital for Children, London
  - Royal Manchester Childrens Hospital, Manchester
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brincidofovir | Standard of Care
Started | 20 | 9
Completed | 11 | 5
Not Completed | 9 | 4
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Study terminated | 4 | 3
Not completed — Investigator Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Due to the premature termination of this study, statistical analyses were not performed. Limited demographic, efficacy, and safety data are provided for the 29 subjects who were enrolled as descriptive summaries.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brincidofovir | Standard of Care | Total
Number analyzed (Participants) | 20 | 9 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 9 | 29
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.1 (4.05) | 5.9 (4.18) | 5.3 (4.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 12 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 18 | 8 | 26
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 17 | 4 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6
  United Kingdom | 12 | 5 | 17
  Italy | 0 | 1 | 1
  France | 3 | 0 | 3
  Germany | 1 | 1 | 2
Adenovirus in plasma [Count of Participants; unit: Participants] — Subjects must have had qualifying adenovirus (AdV) viremia within 100 days of transplant, which was defined as either (1) confirmed AdV viremia of ≥1000 copies/mL and rising on 2 consecutive adenovirus DNA polymerase chain reaction (PCR) tests results (drawn at least 48 hours apart) from the designated central virology laboratory, with the second result being greater than the first; or (2) a single AdV viremia result of ≥10,000 copies/mL from the designated central virology laboratory.
  Participants | 20 | 9 | 29

OUTCOME MEASURES:

1. Primary Outcome: Time-averaged Area Under the Concentration-time Curve for Plasma Adenovirus Viremia (Log10 Copies/mL).
Description: The primary efficacy endpoint for this study was the time-averaged area under the concentration-time curve for plasma adenovirus (AdV) viremia (log10 copies/mL) from randomization through Week 16 post-randomization. Due to the small number of subjects enrolled in the study, formal efficacy analyses were not performed. Individual subject AdV viremia profiles show the differential anti-adenoviral effect of brincidofovir (BCV) in comparison to standard of care (SoC) therapy.
Time Frame: From randomization to 16 weeks post-randomization
Population: The time-averaged area under the concentration-time curve for plasma adenovirus (AdV) viremia was not calculated because many of the viral response data were arbitrarily truncated/censored and individual subject AdV viremia profiles cannot be reported due to concerns with patient confidentiality.
Arm/Group | Brincidofovir | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization to 16 weeks post-randomization.
Description: Note: Other Adverse Events includes non-serious and serious adverse events.
Arm/Group | Brincidofovir | Standard of Care
All-Cause Mortality (participants affected / at risk) | 4/20 | 1/9
Serious Adverse Events (participants affected / at risk) | 15/20 | 6/9
Other Adverse Events (participants affected / at risk) | 20/20 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brincidofovir (N=20) | Standard of Care (N=9)
Evans Syndrome (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 3
Unevaluable event (Gastrointestinal disorders) | 1 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 0
Adenovirus infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 2 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Astrovirus test positive (Investigations) | 1 | 0
Blood creatinine abnormal (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brincidofovir (N=20) | Standard of Care (N=9)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Evans Syndrome (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Thrombotic microanglopathy (Blood and lymphatic system disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 6 | 1
Mucosal inflammation (General disorders) | 1 | 1
Pyrexia (General disorders) | 8 | 5
Venoocclusive liver disease (Hepatobiliary disorders) | 2 | 0
Engraftment syndrome (Immune system disorders) | 2 | 0
Graft versus host disease (Immune system disorders) | 0 | 2
Graft versus host disease in skin (Immune system disorders) | 2 | 2
Adenovirus infection (Infections and infestations) | 3 | 0
Device related infection (Infections and infestations) | 2 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 2
Rhinovirus infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 1 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Fluid balance positive (Investigations) | 0 | 1
Gamma-glutamyltranferase increased (Investigations) | 4 | 2
Haemoglobin decreased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 1
Liver function test increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The study was terminated in May 2019 due to poor subject accrual rates. As a result, statistical analyses were not performed. Limited demographic, efficacy, and safety data are provided for the 29 subjects who were enrolled as descriptive summaries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 12 months after the end of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given opportunity to review and comment. Institution publication may be delayed up to an additional 3 months to allow Sponsor to seek patent protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT03339401/Prot_SAP_003.pdf